CLINICAL TRIAL: NCT02898961
Title: Impact of 30 mg/kg Amikacin and 8 mg/kg Gentamicin on Serum Concentrations in Critically Ill Patients With Severe Sepsis
Acronym: Aminoside_II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2015/JYL-01
Record Dates: First submitted 2016-09-01; First posted 2016-09-13 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2020-12

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Amikacin; Gentamicins

ARMS (1):
- The study population (Experimental): ICU patients with severe sepsis treated with aminoglycosides were recruited.
  Intervention: 30 mg/kg amikacin or 8 mg/kg gentamicin
  Interventions: Drug: 30 mg/kg amikacin or 8 mg/kg gentamicin

INTERVENTIONS:
Drug: 30 mg/kg amikacin or 8 mg/kg gentamicin — In order to improve the achievement of target peak concentrations, either 30 mg/kg amikacin or 8 mg/kg gentamicin was prescribed in ICU patients with severe sepsis.
  In combination with broad-spectrum antibiotics, according to the suspected pathogens and local clinical practice, 30 mg/kg amikacin or 8 mg/kg gentamicin was given (30 min intravenous infusion; the dosage ampoule was systematically emptied with a 5 ml flush). The peak serum concentration sampling occurred 30 minutes after the end of the infusion.

SUMMARY:
Low first-dose peak serum concentrations of amikacin and gentamicin are commonly reported in ICU patients. The present study aimed to assess whether 30 mg/kg amikacin or 8 mg/kg gentamicin achieved target concentrations in ICU patients with severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* ICU patient with severe sepsis
* Treated with aminoglycosides

Exclusion Criteria:

* Renal replacement therapy
* Allergy to aminoglycosides
* Confirmed and/or suspected to have myasthenia
* ICU-acquired neuromuscular disorder
* Under guardianship
* Prisoners
* The patient has already participated in the present protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Presence/absence of target peak serum concentration of aminosides | 30 minutes after the end of the infusion.
  Achievement of targeted peak serum concentration?

REFERENCES:
- [Result] Roger C, Nucci B, Louart B, Friggeri A, Knani H, Evrard A, Lavigne JP, Allaouchiche B, Lefrant JY, Roberts JA, Muller L. Impact of 30 mg/kg amikacin and 8 mg/kg gentamicin on serum concentrations in critically ill patients with severe sepsis. J Antimicrob Chemother. 2016 Jan;71(1):208-12. doi: 10.1093/jac/dkv291. Epub 2015 Oct 1. PMID 26429564